CLINICAL TRIAL: NCT03141697
Title: Is CO2 Insufflation an Amelioration of Routine Colonoscopy?
Brief Title: The Use of CO2 in Routine-Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Juergen Feisthammel, Medical Doctor, Principal Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CO2 Colonoscopy
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Colonoscopy
Keywords: Carbon Dioxide; Coloboscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbon Dioxide (Experimental): Colonoscopy with Insufflation of Carbon Dioxide
  Interventions: Device: Carbon Dioxide
- Room Air (Placebo Comparator): Colonoscopy with Insufflatioin of Room Air
  Interventions: Device: Room air

INTERVENTIONS:
Device: Carbon Dioxide — Insufflation of Carbon Dioxide
  Arms: Carbon Dioxide
Device: Room air — Insufflation of room air
  Arms: Room Air

SUMMARY:
In this double-blind, randomised and controlled study 150 Patients referred to colonoscopy were assigned to either CO2 or air insufflation. We recorded basic characteristics of colonoscopy and the amount of drugs used for sedation. Patients and investigators filled out questionnaires to record pain, abdominal bloating and flatulence.

DETAILED DESCRIPTION:
Between April 2012 and August 2014 150 patients referred to the University Hospital of Leipzig for colonoscopy were randomly assigned to either CO2 or air insufflation.

All examinations were performed by one of four experienced endoscopists. The patients usually received sedation. For sedation midazolam and propofol was used. At the beginning of the examination the patients usually received between 3-5 mg of midazolam and 20-40 mg propofol. During endoscopy propofol was titrated by administration of 20 mg at the time according to and pain reaction of the patient and required depth of sedation.

All patients had nasal insufflation of oxygen with 2 litres per minute. All sedated patients were monitored for pulse, blood pressure and blood oxygen saturation.

For bowel cleansing a solution of Macrogol 3350 (Moviprep®, Norgine) was administered orally according to the manufacturer.

All colonoscopies were performed using Fujifilm Endoscopes (EC 590 Series). For examinations with use of carbon dioxide the Fujifilm CO2 Insufflator GW-1 was used with appropriate water bottle and endoscope valve. The air pump of the light source Fujifilm System 4400 was deactivated according to the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* informed consent

Exclusion Criteria:

* former colonic resections
* severe heart or lung disease (NYHA III or IV)
* Pregnancy
* Patients with planned gastroscopy within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Post-procedural pain | 0 - 24 hrs after colonoscopy
  Pain after Colonoscopy, assessed by visual analog scale (VAS)

SECONDARY OUTCOMES:
Abdominal bloating | 0 - 24 hrs after colonoscopy
  Abdominal bloating, assessed by questionaire
flatulence | 0 - 24 hrs after colonoscopy
  flatulence, assessed by questionaire
procedure time | duration of colonoscopy
  time used for colonoscopy
Used amount of sedative drugs | during endoscopy
  Amount of midazolam and propofol administrated during colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided